CLINICAL TRIAL: NCT05435820
Title: Near-infrared Transcranial Laser Therapy in Subjects With Major Depressive Disorder: A Study of Dosing With Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peruvian Clinical Research (Other)
Collaborators: NeuroThera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NITLT01
Record Dates: First submitted 2022-06-08; First posted 2022-06-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder
Keywords: Near-infrared transcranial laser therapy; Hamilton Depression rating scale; Major depressive Disorder; Clinical trial
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- BCW group (Experimental): NIR-TLT dose:
  i. Treatment site(s): EEG F3 and F4 ii. Temporal format: continuous wave iii. Average radiance: 350 mW / cm2 iv. Exposure time: 429 sec. v. Total fluence delivered: 3.6 kJ (1.8 kJ per treatment location)
  Interventions: Device: Near-infrared Transcranial Laser Therapy
- BPW-1 group (Experimental): NIR-TLT dose:
  i. Treatment site(s): EEG F3 and F4 ii. Temporal format: pulsed wave, 10 Hz; 50% duty cycle iii. Average radiance: 350 mW / cm2 iv. Exposure time: 429 sec. v. Total fluence delivered: 3.6 kJ (1.8 kJ per treatment location)
  Interventions: Device: Near-infrared Transcranial Laser Therapy
- BPW-2 group (Experimental): NIR-TLT dose:
  i. Treatment site(s): EEG F3 and F4 ii. Temporal format: pulsed wave, 40-50 Hz; 50% duty cycle iii. Average radiance: 350 mW / cm2 iv. Exposure time: 429 sec. v. Total fluence delivered: 3.6 kJ (1.8 kJ per treatment location)
  Interventions: Device: Near-infrared Transcranial Laser Therapy
- SHAM group (Sham Comparator): NIR-TLT dose:
  i. Treatment site(s): none ii. Temporal format: none iii. Average radiance: 0 mW / cm2 iv. Exposure time: 429 sec. v. Total fluence delivered: 0 kJ
  Interventions: Device: Near-infrared Transcranial Laser Therapy

INTERVENTIONS:
Device: Near-infrared Transcranial Laser Therapy — The treatment consists in exposing bilaterally the frontal brain to Transcranial Laser Therapy, which may enhance ATP production in depressed subjects.

SUMMARY:
The Near-infrared transcranial laser therapy (NIR-TLT) is a non-ionizing electromagnetic wave. The NIR-TLT is invisible, penetrates the skin and skull into brain tissue and is non-invasive. The benefits of NIR-TLT are wavelength specific. A mitochondrial enzyme, the Cytochrome c oxidase, is the primary chromophore for the NIR-TLT with a wavelength of around 830 nm. When this enzyme is activated, it leads to increased adenosine triphosphate (ATP) production and this event is related to the promotion of cellular plasticity and cytoprotection. These are critical cellular processes for recovery of the depressive patients. Therefore, this study will contribute to answer the question of whether NIR-TLT has an antidepressant effect and whether it is acceptable in minority population.

DETAILED DESCRIPTION:
Study purpose: The main aim is to assess and compare the effect(s) of each of the four doses of the Near-infrared Transcranial Laser Therapy (NIR-TLT) on the symptomatology of depression: antidepressant effect, in subjects with major depressive disorder (MDD). Study design: This protocol is a multicentered, randomized, simulated, and double-blind clinical study. This work will randomize 112 subjects into 4 equal groups: bilateral continuous wave (BCW), bilateral pulsed wave (BPW 1-2) y SHAM. All subjects, investigators (except the study statistician), and outcomes assessors will be blind to group assignment. The device operator will be aware of group assignments. All subjects will receive 3 NIR-TLT treatments per week for 6 weeks. A follow-up evaluation will be performed 2 weeks after the end of the study. The treatment will follow these specifications: wavelength 830 nm; average irradiance 54,8 mW / cm2; average fluence of 65,8 J / cm2 (consistently with parameters used in the ELATED-2 study at MGH with the device Omnilux New U), being the total Fluency delivered: 3.6 kJ (bilateral) o 1.8 kJ (unilateral), either on the subject's forehead, at or near electroencephalography sites (EEG) F3 and F4. All NIR-TLT sessions will last 20 minutes, regardless of group assignment. Study population: Patients eligible for study participation will be diagnosed with major depressive disorder (MDD) by DSM criteria. Subjects will be between 18-75 years of age (have not had 76st birthday) on the date of screening. Duration of participation: Subjects will be followed in the study for 8 weeks (a 6-week treatment period, plus 2 weeks of follow-up). The total duration of the study will be 24 months. Assessment criteria: The primary efficacy criteria is the improvement in depressive symptoms from each of the four doses of NIR-TLT. Assessed using HAMD-17, at 3 time points (visit 1, visit 9 and visit 18).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age at screening will be between 18 and 75 years old (inclusive).
2. Diagnosis of major depressive disorder (Mini International Neuropsychiatric Interview, MINI)
3. QIDS-CR≥12 at screening
4. CGI-S ≥4 or higher, i.e., "moderately depressed"
5. Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms plus spermicide) if sexually active.
6. Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
7. The subject is willing to participate in this study for at least 12 weeks.
8. Subjects will need to be on stable dose(s) of antidepressants (if taking any) for at least six weeks prior to enrollment.

Exclusion Criteria:

1. Decrease in Symptoms of Depression Questionnaire (SDQ) self-report from screening to baseline >=30%, calculated as [(SDQ screening-88) - (SDQ initial-88) / (SDQ screening-88)] >=30/100. A score of 88 is "normal" in SDQ.
2. The subject is pregnant or lactating.
3. The subject failed more than 2 adequate treatments with FDA approved antidepressants during current episode per Antidepressant Treatment Response Questionnaire (ATRQ) criteria (less than 50% decrease in depressive symptomatology).
4. Structured psychotherapy focused on treating the subject's depression is permitted if started at least 8 weeks prior to the screening visit.
5. Substance dependence or abuse in the past 3 months.
6. History of a psychotic disorder or psychotic episode (current psychotic episode per MINI assessment).
7. Bipolar affective disorder (per MINI assessment).
8. Unstable medical illness, defined as any medical illness which is not well-controlled with standard-of-care medications (e.g., insulin for diabetes mellitus).
9. Active suicidal or homicidal ideation (both intention and plan are present), as determined by Columbia-Suicide Severity Rating Scale (C-SSRS) screening.
10. The subject has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that is found to be in proximity to any of the procedure sites.
11. The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, implantable shunt - Hakim valve).
12. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudine (verteporfin) for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer)
13. Recent history of stroke (90 days).
14. The subject failed a device-based intervention FDA-approved for the treatment of depression, during the current episode (e.g. less than 50% decrease in depressive symptomatology with Transcranial Magnetic Stimulation).
15. History of dementia, traumatic brain injury (TBI) or any other organic neurological disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Changes in the scores of the Hamilton Depression Rating Scale (HAMD-17) from baseline to week 3 and week 6. | From baseline to week 3 and week 6.
  The antidepressant effects of NIR-TLT doses will be measured using the Hamilton Depression rating scale (HAM-D 17). The HAM-D 17 is a 17-item clinician rated instrument developed to quantify the severity of depression in subjects already diagnosed with this disorder. The rating of this tool will be determined in an interview with the psychiatrist, yielding a maximum score of 52. Higher scores represent greater severity of depression.

SECONDARY OUTCOMES:
Changes in the scores of the Quick Inventory of Depressive Symptomatology-Clinician Rated Scale (QIDS-CR) from baseline to week 3 and week 6. | From baseline to week 3 and week 6.
  The antidepressant effects of NIR-TLT doses will be measured using the QIDS-CR. This is a brief (16-item) clinician-rated inventory of core depressive symptoms such as sleep, depressed mood, appetite, concentration, suicidal ideation, interest, energy, psychomotor retardation, or agitation. The range score is 0 to 27. Higher scores represent greater severity of depression.
Changes in the scores of the Clinical Global Impressions - Severity (CGI-S) from baseline to week 3 and week 6. | From baseline to week 3 and week 6.
  The antidepressant effects of NIR-TLT doses will be measured using the CGI-S. The CGI-S is one of the two components of the CGI test. This tool asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Changes of electroencephalogram (EEG) espectral power from baseline to week 3 and week 6. | From baseline to week 3 and week 6.
  To compare the effects of NIR-TLT doses on brain electrophysiology, changes in EEG spectral power in all spectral bands for each dose will be analyzed. The waves that will be considered are alpha, theta, and delta. For all of them, frequency and amplitude will be registered.
Changes in the scores of the Systemic Assessment for Treatment Emergent Events (SAFTEE-SI) from baseline to week 3 and week 6. | From baseline to week 3 and week 6.
  To compare the safety and tolerability of NIR-TLT doses, mean changes in SAFTEE-SI scores will be analyzed. This is a questionnaire developed for psychiatric trials. The SAFTEE-SI allows ratings of five levels of severity and collects information about the onset, duration, pattern, judgment of attribution of cause, and action taken by the clinician when an Adverse Event happens. The range score is 0 to 128.
Brain metabolism effect of NIR-TLT dose (exploratory assessment) from baseline to week 6. | From baseline to week 6.
  The analysis of the results obtained in the PET will be for exploratory purposes to study the brain metabolism of the participants, before and at the end of the study intervention in the 4 groups. The cortical regions that will be analyzed are the prefrontal lateral and prefrontal medial regions (right and left for both).

CONTACTS AND LOCATIONS:
Overall Officials: William Aguilar Rivera, Dr., Principal Investigator — Hospital Nacional Hipolito Unanue; Beatrice Macciotta Felices, Dr., Principal Investigator — Clinica Vesalio
Locations (1):
- Hospital Nacional Hipolito Unanue, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
After the completion of the study, the researchers will decide if IPDs can be shared. The data will first be sent to the regulatory institutions involved.

REFERENCES:
- [Background] Cassano P, Petrie SR, Mischoulon D, Cusin C, Katnani H, Yeung A, De Taboada L, Archibald A, Bui E, Baer L, Chang T, Chen J, Pedrelli P, Fisher L, Farabaugh A, Hamblin MR, Alpert JE, Fava M, Iosifescu DV. Transcranial Photobiomodulation for the Treatment of Major Depressive Disorder. The ELATED-2 Pilot Trial. Photomed Laser Surg. 2018 Dec;36(12):634-646. doi: 10.1089/pho.2018.4490. Epub 2018 Oct 20. PMID 30346890
- [Background] Cassano P, Cusin C, Mischoulon D, Hamblin MR, De Taboada L, Pisoni A, Chang T, Yeung A, Ionescu DF, Petrie SR, Nierenberg AA, Fava M, Iosifescu DV. Near-Infrared Transcranial Radiation for Major Depressive Disorder: Proof of Concept Study. Psychiatry J. 2015;2015:352979. doi: 10.1155/2015/352979. Epub 2015 Aug 19. PMID 26356811
- [Background] Caldieraro MA, Cassano P. Transcranial and systemic photobiomodulation for major depressive disorder: A systematic review of efficacy, tolerability and biological mechanisms. J Affect Disord. 2019 Jan 15;243:262-273. doi: 10.1016/j.jad.2018.09.048. Epub 2018 Sep 17. PMID 30248638